CLINICAL TRIAL: NCT05949957
Title: Harnessing Human Potential and Improving Health Span in Women and Their Children: a Randomized Controlled Trial and Follow-up (HAPPY STUDY)
Brief Title: Harnessing Human Potential and Improving Health Span in Women and Their Children
Acronym: HAPPY
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institute for Human Development and Potential (IHDP), Singapore (Other)
Responsible Party: Principal Investigator, Johan Eriksson, Senior Principal Investigator, Institute for Human Development and Potential (IHDP), Singapore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2023/00178; 2023/00178 (Other: Singapore Institute for Clinical Sciences (SICS))
Record Dates: First submitted 2023-06-08; First posted 2023-07-18 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Type 2 Diabetes; Healthy Lifestyle Behaviors; Gestational Diabetes
Keywords: Type 2 Diabetes; Gestational Diabetes Mellitus; Women; Prevention; Healthy lifestyle; Physical activity; Diet; Sleep; Mental wellbeing; Digital health interventions
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes, Gestational; Motor Activity

STUDY DESIGN:
Intervention Model Description: A parallel 2-arm, single-Centre Randomized Control Trial based on 1:1 allocation ratio. Eligible women will be randomized at baseline to either Group 1 (Intervention) or Group 2 (Control). Participants will receive the assigned intervention from baseline to 1 year, followed by 3 years follow-up period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): LvL UP App (Smarphone-based conversational agent-delivered holistic lifestyle intervention for the prevention of type 2 diabetes, and common mental disorders [anxiety, depression]).
  HAPPY App (Health promotion information, and display health data collected)
  Oura ring and Oura App (activity-tracking wearable that collects lifestyle data [physical activity, sleep and heart rate]).
  Interventions: Behavioral: LvL UP App; Behavioral: HAPPY App; Behavioral: Oura Ring And Oura App
- Control group (Active Comparator): HAPPY App (Health promotion information, and display health data collected)
  Oura ring and Oura App (activity-tracking wearable that collects lifestyle data [physical activity, sleep and heart rate]).
  Interventions: Behavioral: HAPPY App; Behavioral: Oura Ring And Oura App

INTERVENTIONS:
Behavioral: LvL UP App — LvL UP App: A Smartphone-based conversational agent-delivered holistic lifestyle intervention. The intervention group will receive several digital coaching sessions focus on 3 pillars: diet, physical activity, and mental well-being to promote health literacy and promote healthy lifestyles. The app includes practical exercises per pillar (e.g., journaling, slow-breathing exercises, lifehacks).
  Arms: Intervention group
Behavioral: HAPPY App — HAPPY App: Each subject will use the HAPPY App that aims to:(1) deliver health promotion information (guided by Singapore Health Promotion Board's resources), and (2) display health data collected (e.g., body mass index, blood pressure, OGTT results) that help them monitor own health and prevent T2D.
Behavioral: Oura Ring And Oura App — Oura ring and Oura App: Each subject will receive an Oura ring, i.e., an activity-tracking wearable that collects lifestyle data (physical activity, sleep and heart rate (as a proxy for stress) that will be synced with Oura App

SUMMARY:
Women with Gestational Diabetes Mellitus (GDM) are 12-times more likely to develop Type 2 Diabetes (T2D) 4-6 years after delivery than women without GDM. There has been evidence that lifestyle modifications such as physical activity (PA), dietary intake, sleep, and stress management can prevent or delay type 2 diabetes (T2D). The purpose of this study is to assess the efficacy of a holistic lifestyle digital health intervention with post-GDM women in large community settings in Singapore. The study consists of a 1-year randomized controlled trial (RCT) with 3 years follow-up. Women who are eligible for the study will be randomized to either Group 1 (Intervention) or Group 2 (Control) at baseline. Both groups will be followed in years 2-4. Women from both groups will be provided with an Oura ring for tracking physical activity, sleep, and heart rate variability (a proxy for stress), and the "HAPPY app," which will provide health promotion information about physical activity, diet, sleep, and mental wellbeing, as well as display the information collected (such as body mass index, blood pressure, and OGTT results). The active group will receive the "LVL UP app" a smartphone-based chatbot-delivered intervention, designed to provide personalized recommendations through multiple digital coaching sessions aimed at improving health literacy and practicing healthy lifestyles to prevent Type 2 diabetes and common mental disorders (i.e., anxiety, depression).

DETAILED DESCRIPTION:
The overall goal of this study is to reduce the risk of Type 2 diabetes (T2D) and pre-diabetes in Asian women and their children by focusing upon a major high-risk group - women with a history of gestational diabetes (GDM) in Singapore. GDM is diabetes diagnosed for the first-time during pregnancy and has traditionally been considered a benign condition because typically glucose levels return to normal after delivery. Women with pregnancies complicated by GDM often progress to develop T2D later in life.

There is evidence that holistic lifestyle modifications that include strategies to improve dietary intake, physical activity, and mental well-being can prevent or delay the onset of type 2 diabetes. The use of digital health interventions can also assist in the prevention of T2D. However, limited studies have been conducted with Asian populations.

This study aims (1) to identify post-GDM women from large community settings in Singapore and to assess the efficacy of a holistic lifestyle digital intervention (focusing on diet, physical activity, sleep, and mental well-being) on glucose regulation with those identified women.

Secondary objectives are: (a) to examine the potential impacts of the proposed intervention on the health and well-being of subjects' family members (e.g., children); (b) to determine the diabetes risk of the subjects over a 3-year follow-up period; (c) to explore potential economic impacts of the proposed intervention (e.g., healthcare expenditures); (d) to study the importance of gut microbiota and epigenetic factors in relation to changes in glucose metabolism, and (e) to ascertain the safety of the proposed intervention.

The study is a 1-year randomized controlled trial with three years of follow-up. The primary outcomes involved the incidence of Type 2 diabetes confirmed by a 2-hr 75g Oral Glucose Tolerance Test (OGTT) over a 4-year period. Secondary outcomes are (1) incidence of impaired fasting glucose and impaired glucose tolerance; (b) changes in cardiometabolic variables (e.g., body weight, HbA1c, insulin, blood lipids, blood pressures) in the women; (c) changes in women's body composition; (d) changes in women's mental well-being (e.g., defined by BDI-II, STAI, WHO-5, PSS-4); (e) changes in the health and wellbeing of their children, and (f) a composite of major adverse events (MAE) comprising fatal and non-fatal events associated with Type 2 diabetes.

Eligible women will be randomized at baseline to either Group 1 (Intervention) or Group 2 (Control) for 1 year.

Group 1 (Intervention) consists of several virtual coaching sessions about healthy lifestyle delivered by a conversational agent (chatbot) embedded in the LvL UP App within 24 weeks (weeks 2 to 26) to complete three levels of health literacy. Additionally, individuals will receive an Oura ring at baseline (activity-tracking wearable that collects lifestyle data), as well as the HAPPY App (educational content about lifestyle and health outcomes [e.g., body mass index, blood pressure, OGTT results]).

Group 2 (Control) subjects will receive an Oura ring at baseline, and the HAPPY App

Follow-up Period Upon completion of the one-year RCT period, both groups will be followed-up for 3 years. During the follow-up visits, body measurements, OGTT, bio-sampling, and data collection will be conducted.

Both groups will be assessed at baseline, week 26, 1 year visit, 2-year visit (follow-up 1), 3-year visit (follow-up 2), and 4-year visit (follow-up 3)

ELIGIBILITY:
Inclusion Criteria:

1. Female, age: 21 - 45 years
2. Had a history of GDM (at least 1 year and not more than 10 years)
3. Chinese, Malay or Indian ethnic groups
4. Body mass index (at least 18.5 kg/m2 and not more than 35 kg/m2)
5. Not planning to conceive in the next one year
6. Not performing exclusive breastfeeding during study period
7. Own a smartphone compatible with the study mobile Apps
8. Proficient in English language
9. Plan to stay in Singapore for the next 4 years
10. Willing to comply to study protocol
11. Able to provide a written informed consent

Exclusion Criteria:

1. Current or previous diagnosis of diabetes (Type 1 or 2), except GDM
2. Currently pregnant
3. Given birth within the last 12 weeks
4. Severely limited mobility (e.g., wheelchair bound, require long-term walking aid, etc.)
5. Diagnosed with malnutrition or eating disorder
6. Diagnosed with cancers, unstable heart diseases, severe kidney diseases, severe liver diseases
7. Diagnosed with severe insomnia, unstable mental conditions, dementia, or cognitive impairment
8. Experienced alcohol or drug abuse
9. Currently having medications known to influence glucose metabolism (e.g. peroral corticosteroids)
10. Currently participating in concurrent clinical trial or lifestyle intervention study

Ages: 21 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 400 (Estimated)
Dates: Start 2023-10-20 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Glucose Tolerance Changes | Changes in glucose over four years, including: Baseline, Year1, Year 2 (Follow-up 1), Year 3(Follow-up 2), Year 4(Follow-up 3)
  2-hr 75g Oral Glucose Tolerance Test (OGTT)

SECONDARY OUTCOMES:
Anthropometric Measurements | Baseline, Week 26/27 (Midpoint Visit), Year1, Year 2 (Follow-up 1), Year 3(Follow-up 2), Year 4(Follow-up 3)
  Participants will be measured for their height in feet and weight in kilograms. Weight and height will be combined to report BMI in kg/m^2.
Blood pressure (BP) | Baseline, Week 26 (Midpoint Visit), Year1, Year 2 (Follow-up 1), Year 3(Follow-up 2), Year 4(Follow-up 3)
  Blood pressure will be measured using an automated blood pressure monitor.
Biosample Collection (Fasting blood) | Baseline, Week 26 (Midpoint Visit), Year1, Year 2 (Follow-up 1), Year 3(Follow-up 2), Year 4(Follow-up 3)
  Fasting blood draw will be analyzed for HbA1c & fasting blood glucose
Biosample Collection (Saliva) | Baseline, Week 26 (Midpoint Visit), Year1, Year 2 (Follow-up 1), Year 3(Follow-up 2), Year 4(Follow-up 3)
  Saliva collected using Salivette® kit (cortisol)
Biosample Collection (Buccal swab) | Baseline, Week 26 (Midpoint Visit), Year1, Year 2 (Follow-up 1), Year 3(Follow-up 2), Year 4(Follow-up 3)
  Buccal swab collected using Isohelix kit (DNA profiling)
Biosample Collection (Stool) | Baseline, Week 26 (Midpoint Visit), Year1, Year 2 (Follow-up 1), Year 3(Follow-up 2), Year 4(Follow-up 3)
  Stool collected via OMNIgene®•GUT OM-200 (Gut microbiota)
Bioelectrical Impedance Analysis (BIA) | Baseline, Week 26 (Midpoint Visit), Year1, Year 2 (Follow-up 1), Year 3(Follow-up 2), Year 4(Follow-up 3)
  BIA is a non-invasive technology that can accurately measure a person's total body water, extracellular and intracellular fluid volumes.
Depression | Baseline, Week 26 (Midpoint Visit), Year1, Year 2 (Follow-up 1), Year 3(Follow-up 2), Year 4(Follow-up 3)
  Beck Depression Inventory II (BDI-II)
Anxiety | Baseline, Week 26 (Midpoint Visit), Year1, Year 2 (Follow-up 1), Year 3(Follow-up 2), Year 4(Follow-up 3)
  The State-Trait Anxiety Inventory (STAI)
Health Status | Baseline, Week 26 (Midpoint Visit), Year1, Year 2 (Follow-up 1), Year 3(Follow-up 2), Year 4(Follow-up 3)
  The Short Form (36) Health Survey (SF-36)
Sleep | Baseline, Week 26 (Midpoint Visit), Year1, Year 2 (Follow-up 1), Year 3(Follow-up 2), Year 4(Follow-up 3)
  PSQI: The Pittsburgh Sleep Quality Index (PSQI
Lifestyle | Baseline, Year1, Year 2 (Follow-up 1), Year 3(Follow-up 2), Year 4(Follow-up 3)
  e-Diary (Qualtrics survey system) self-report lifestyle
Social-emotional development (Children) | Baseline, Year1, Year 2 (Follow-up 1), Year 3(Follow-up 2), Year 4(Follow-up 3)
  ASQ:-3: Ages and stages questionnaire: social-emotional development screening tool is used to assess children's (for age 2 month - 60 months) self-regulation, communication, autonomy, compliance, adaptive functioning, affect, and interaction with people.

OTHER OUTCOMES:
Cognitive emotion regulation strategies | Baseline, Week 26 (Midpoint Visit), Year1
  CERQ: Cognitive Emotion Regulation Questionnaire
Sleep wake up | Baseline, Week 26 (Midpoint Visit), Year1
  MEQ:The morningness-eveningness questionnaire
Happiness | Baseline, Week 26 (Midpoint Visit), Year1
  SHS: Subjective Happiness Scale
Health Literacy | Baseline, Week 26 (Midpoint Visit), Year1
  HLQ: Health Literacy Questionnaire
Stress | Baseline, Week 26 (Midpoint Visit), Year1
  PSS-4: Perceived Stress Scale 4
Mental Wellbeing | Baseline, Week 26 (Midpoint Visit), Year1
  WHO-5 wellbeing Index
Infant sleep | Baseline, year 1
  BISQ-R-SF: Brief infant sleep questionnaire is on parent-reported toddler (0-3 years) sleep over prior 1 week.
Child and Mother Interaction | 12 months (Year 1 visit)
  StimQ-toddler (for age 1-3 years) / StimQ-pre-school (for age 4-5 years) is designed to find out the different types of toys and games that mothers have for child in the home, and the kinds of activities that mother and child do together.
Child's Sleep Habits | Baseline, year 1
  CSHQ: Child's Sleep Habits Questionnaire (for age 4-5 years) assesses the frequency of children behaviors associated with common pediatric sleep difficulties.

CONTACTS AND LOCATIONS:
Locations (1):
- Singapore Institute for Clinical Sciences (SICS), Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Salamanca-Sanabria A, Liew SJ, Mair J, De Iorio M, Ling YDY, Tint MT, Wei YT, Lim K, Ong D, Chooi YC, Tay V, Eriksson JG. A holistic lifestyle mobile health intervention for the prevention of type 2 diabetes and common mental disorders in Asian women with a history of gestational diabetes: a randomised control trial with 3-year follow-up protocol. Trials. 2024 Jul 3;25(1):443. doi: 10.1186/s13063-024-08247-x. PMID 38961430